CLINICAL TRIAL: NCT01802840
Title: Soy Fiber Improves Weight Loss And Lipid Profile In Overweight And Obese Adults: A Randomized Controlled Trial
Brief Title: Soy Fiber Improves Weight Loss and Lipid Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Xiaojie Hu, Msd, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 12-01
Record Dates: First submitted 2013-02-23; First posted 2013-03-01 (Estimated); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Obesity; Overweight; Weight Loss
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- biscuits without soy fiber (Placebo Comparator): biscuits without soy fiber
  Interventions: Dietary Supplement: biscuits supplemented with soy fiber
- biscuits supplemented with soy fiber (Experimental): biscuits supplemented with soy fiber
  Interventions: Dietary Supplement: biscuits supplemented with soy fiber

INTERVENTIONS:
Dietary Supplement: biscuits supplemented with soy fiber — Thirty nine overweight and obese college adults (19-39 y of age) were randomly assigned to consume control biscuits or biscuits supplemented with soy fiber for 12 wk (approximately 100g/d).

SUMMARY:
The aim of this study is to examine the effects of soy fiber on body weight, body composition and blood lipids in overweight and obese participants.

DETAILED DESCRIPTION:
Thirty nine overweight and obese college adults (19-39 y of age) were randomly assigned to consume control biscuits or biscuits supplemented with soy fiber for 12 wk (approximately 100g/d). Information on body weight, body mass index, waist/hip circumference, blood pressure as well as measures of lipoprotein, glucose concentrations, and HbA1c was obtained at baseline, 8 and 12 wk after intervention. Body composition was also assessed at baseline and wk 12, respectively.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 23-35 kg/m2

Exclusion Criteria:

* Subjects taking any drugs, botanicals or nutraceutical known to influence body weight or blood pressure
* significant history of eating disorders
* strenuous exercise to lose weight
* lipid-lowering medication
* use of steroids and other agents that may influence lipid metabolism
* hyperlipidemia
* hyperglycemia
* diabetes mellitus
* cardiovascular disease
* major systemic diseases
* gastrointestinal problems
* liver and renal failure

Ages: 19 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
weight loss | 12 weeks
  Body weight of participants in soy fiber group was decreased significantly over the study period compared with the baseline.

SECONDARY OUTCOMES:
serum levels of total cholesterol | 12 weeks
  Serum levels of total cholesterol of participants in soy fiber group was decreased significantly over the study period compared with the baseline.
serum levels of low density lipoprotein cholesterol | 12 weeks
  Serum levels of low density lipoprotein cholesterol of participants in soy fiber group was decreased significantly over the study period compared with the baseline.
body fat | 12 weeks
  Body fat of participants in soy fiber group was lowered significantly at wk 12 than that of baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Duo Li, Prof., Study Director — Zhejiang University
Locations (1):
- Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Maki KC, Beiseigel JM, Jonnalagadda SS, Gugger CK, Reeves MS, Farmer MV, Kaden VN, Rains TM. Whole-grain ready-to-eat oat cereal, as part of a dietary program for weight loss, reduces low-density lipoprotein cholesterol in adults with overweight and obesity more than a dietary program including low-fiber control foods. J Am Diet Assoc. 2010 Feb;110(2):205-14. doi: 10.1016/j.jada.2009.10.037. PMID 20102847
- [Background] Ludwig DS, Pereira MA, Kroenke CH, Hilner JE, Van Horn L, Slattery ML, Jacobs DR Jr. Dietary fiber, weight gain, and cardiovascular disease risk factors in young adults. JAMA. 1999 Oct 27;282(16):1539-46. doi: 10.1001/jama.282.16.1539. PMID 10546693
- [Derived] Hu X, Gao J, Zhang Q, Fu Y, Li K, Zhu S, Li D. Soy fiber improves weight loss and lipid profile in overweight and obese adults: a randomized controlled trial. Mol Nutr Food Res. 2013 Dec;57(12):2147-54. doi: 10.1002/mnfr.201300159. Epub 2013 Jul 23. PMID 23881774